CLINICAL TRIAL: NCT03611933
Title: The Effect of Position Change on Vital Signs, Back Pain and, Vascular Complications Following Percutaneous Coronary Intervention
Brief Title: Effects of Position Change After PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, SELDA MERT, Lecturer Dr., Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16214662/050.01.04/85
Record Dates: First submitted 2018-07-09; First posted 2018-08-02 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Percutaneous Coronary Intervention; Coronary Artery Disease
Keywords: Back pain; patient positioning; vascular complications; vital signs
MeSH Terms: conditions — Coronary Artery Disease; Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized-controlled quasi experimental study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (CG) (No Intervention): Patients in the CG were provided with routine nursing care, as practiced in the clinic, including restricted bed rest. For this purpose, patients were given supine position in which the HOB was elevated 15° for 6-10 h; the patient's leg on the of the side of intervention was kept straight.
- Experimental group (EG) (Experimental): Patients in the EG were applied position changes between the first minute and sixth hour. During the initial six hours a supportive, thin pillow, 4 x 40 x 100 cm in size, was placed between the patient's shoulders and gluteals; this reduced the pressure on local tissues and muscle groups.
  Interventions: Other: position change applied at different times

INTERVENTIONS:
Other: position change applied at different times — Time 1 - in the first fifth minute after the procedure supine position in which the HOB was elevated 15° Time 2 - in the first hour low fowler's position were given in which the HOB was elevated 15-30° Time 3 - in the third hour semi high fowler's position were given in which the HOB was elevated 30-45° Time 4 - in the fourth hour left or right lateral position were given in which the HOB was elevated 15° Time 5 - in the fifth hour low fowler's position were given in which the HOB was elevated 15-30° Time 6 - in the sixth hour standard fowler's position were given in which the HOB was elevated 45-60°
  Arms: Experimental group (EG)

SUMMARY:
Aims and objectives: To determine the effect of position change that is applied after percutaneous coronary intervention on vital signs, back pain, and vascular complications.

Background: In order to minimize the post-procedure complications, patients are restricted to prolonged bed rest that is always accompanied by back pain and and hemodynamic instability.

Design: Randomized-controlled quasi experimental study Methods: The study sample chosen for this study included 200 patients who visited a hospital in Turkey between July 2014 and November 2014. Patients were divided into two groups by randomization. Patients in the control group (CG, n = 100) were put in a supine position, in which the head of the bed (HOB) was elevated to 15°, the patient's leg on the side of the intervention was kept straight and immobile; positional change was applied to patients in the experimental group (EG, n = 100).

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is an interventional procedure used to diagnose and treat chronic coronary artery disease. The recommended period of bed rest following a PCI is reported by Rolley et al. (2011) as being 2-4 hours (h). According to evidence-based guidelines in relevant literature, however, the bed rest was reported from 2-24 h; in these instances the supine position (SP) was used, which leads to movement limitation.

Among the patient-care goals during the post-procedural period, sustaining tissue perfusion and heart and vascular system operation, regulating vital signs, reducing pain, and supporting movement are important. According to such a procedure, the nurse's independent role is to provide the safest position for the patient, thereby positively affecting vital signs after PCI and reducing vascular complications and back pain.

Recently, similar nursing studies have reported the effect of position change after PCI on back pain, as well as vascular complications after PCI, the effect of position change on certain vital signs and vascular complications, the effect of position change regarding pain, patient comfort and certain vital signs, and the effect of positional change on intervention pain and all vital signs. Some studies have also looked into the effect of positional changes on back pain, certain vital signs, and vascular complication.

Prolonged bed rest in a SP has become tradition, but it can have negative effects. Comprehensive studies in the existing literature that can be applied to the post-PCI nursing care process-and which study the effect of the most reliable positional change on all vital signs, vascular complications, and, back pain-display a numerical inadequacy. Consequently, the authors intend the current study to be an experimental investigation of the effect of position change on vital signs, vascular complications, and back pain.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* a 6-7 F catheter
* must be able to lie in a supine position (without breathing problems)
* must be in balance hemodynamically

Exclusion Criteria:

* hypotension
* hyperthermia or hypothermia
* no procedure except for PCI
* coagulation disorder
* decompensated heart failure
* diastolic blood pressure (DBP) > 100 mmHg
* systolic blood pressure (SBP) > 180 mmHg
* vascular complications
* the femoral artery damage
* body mass index ≥ 35 kg/m2
* pre-treatment back pain
* vertebral disc disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Respiratory rate (respiratory rate / min.) | The time from the first 5 minutes to the end of the sixth hour from the first 5th minute to the 6th hour after Percutaneous Coronary Intervention
  physiological parameter - rate per minute
body temperature (centigrade degree -°C) | The time from the first 5 minutes to the end of the sixth hour from the first 5th minute to the 6th hour after Percutaneous Coronary Intervention
  physiological parameter - measured with the use of a electronic thermometer
heart rate (min. / pulse) | from the first 5th minute to the 6th hour from the first 5th minute to the 6th hour after Percutaneous Coronary Intervention
  physiological parameter - beats per minute
systolic and diastolic blood pressure (mmHg) | The time from the first 5 minutes to the end of the sixth hour from the first 5th minute to the 6th hour after Percutaneous Coronary Intervention
  physiological parameter - measured with the use of a blood-pressure monitor
back pain | The time from the first 5 minutes to the end of the sixth hour from the first 5th minute to the 6th hour after Percutaneous Coronary Intervention
  Visual Analog Scale (VAS) for pain- score range = 0 - 10. "0" corresponds to "no pain" and "10" indicates "worst pain imaginable".
Bleeding (present or absent) | The time from the first 5 minutes to the end of the sixth hour from the first 5th minute to the 6th hour after Percutaneous Coronary Intervention
  vascular complication:(a) dressing contaminant, (b) pressure required, (c) dressing contaminant + pressure required, and (d) blood transfusion required
hematoma (cm) | The time from the first 5 minutes to the end of the sixth hour from the first 5th minute to the 6th hour after Percutaneous Coronary Intervention
  vascular complication: 5 centimeters (cm) to greater hematoma, major hematoma; Less than 5 cm hematoma, minor hematoma
Ecchymosis | The time from the first 5 minutes to the end of the sixth hour from the first 5th minute to the 6th hour after Percutaneous Coronary Intervention
  vascular complication: blue-violet coloration of the skin as a result of subcutaneous tissue bleeding

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mert Boga S, Oztekin SD. The effect of position change on vital signs, back pain and vascular complications following percutaneous coronary intervention. J Clin Nurs. 2019 Apr;28(7-8):1135-1147. doi: 10.1111/jocn.14704. Epub 2018 Nov 22. PMID 30367542
- See also: Pubmed — http://pubmed.ncbi.nlm.nih.gov/30367542/